CLINICAL TRIAL: NCT05062408
Title: Impact of the Sustained Viral Response on the Natural History Chronic Hepatitis c After Treatment With Direct Action Antivirals
Brief Title: Impact of the Sustained Viral Response of Chronic Hepatitis c After Treatment With Direct Action Antivirals
Acronym: Hepatitis
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-ANT- 2021-01
Record Dates: First submitted 2021-09-13; First posted 2021-09-30 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases: Patients treated with direct-acting antivirals.

SUMMARY:
The purpose of this study is to evaluate the evolution of liver injury with fibrosis data obtained using non-invasive serological markers in patients who achieved SVR after treatment with direct-acting antivirals.

DETAILED DESCRIPTION:
This open study includes patients with chronic hepatitis C who received treatment with the new direct-acting antivirals between November 1, 2014 and December 31, 2017, who achieved a sustained viral response at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic liver disease caused by virus C.
* Have received treatment with the new DAAs between November 1, 2014 and December 1, 2017.
* Patients diagnosed with advanced fibrosis and liver cirrhosis. Advanced fibrosis was defined as a Fibroscan> 10 kPa, an APRI index> 1.5 and / or a FIB-4 index> 3.25. For its part, cirrhosis was defined such as a Fibroscan> 12.5 kPa and / or presence of esophagogastric varices in the endoscopic study and / or data portal hypertension ultrasound.

Exclusion Criteria:

* Coinfection by virus B or HIV.
* Development of HCC before or during treatment.
* Abuse of alcohol intake or addiction to parenteral drugs.
* Liver disease of non-viral etiology (autoimmune, toxic, metabolic).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are patients with chronic hepatitis C who have been treated with direct-acting antivirals between 2014 and 2017. Also patients with fibrosis and liver cirrhosis.
Sampling Method: Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with a progression of liver injury. | Up to 4 weeks
  To assess the evolution of liver injury with fibrosis data in patients who achieved SVR after treatment with direct-acting antivirals.

SECONDARY OUTCOMES:
Identify patients who develop liver-related events (liver decompensation, hepatocellular carcinoma, and death) after achieving sustained viral response. | Up to 4 weeks.
  Development of hepatic decompensation, defined as a patient with ascites, spontaneous bacterial peritonitis (PBR), digestive bleeding of varicose origin, or hepatic encephalopathy at some point in the evolution from SVR until the end of study follow-up.
Rate of risk factors presented by patients. | Up to 4 weeks.
  Identify risk factors in patients who develop liver complications after achieving sustained viral response.
Absence of improvement in non-invasive fibrosis parameters vs the development of liver complications. | Up to 4 weeks.
  To determine if there is a relationship between the absence of improvement in non-invasive fibrosis parameters and the development of liver complications.
Clinical and fibrosis data. | Up to 4 weeks.
  To compare the clinical and fibrosis data between patients who develop liver complications and those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernández Álvarez, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen macarena, Seville, Spain